CLINICAL TRIAL: NCT03950765
Title: Real-time Intervention for Suicide Risk Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harvard University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Evan Kleiman, Principal Investigator, Harvard University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-1813; R34MH113757-01A1 (NIH)
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Suicide, Attempted; Suicide and Self-harm
Keywords: ecological momentary assessment; ecological momentary intervention; distress
MeSH Terms: conditions — Suicide, Attempted; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ecological Momentary Intervention (Experimental): This group will receive three intervention prompts and three assessment prompts on their smartphone each day.
  Interventions: Behavioral: Ecological momentary intervention

INTERVENTIONS:
Behavioral: Ecological momentary intervention — Content of this intervention is based on pre-established transdiagnostic protocols for addressing the negative emotion associated with suicidal thoughts and behaviors.

SUMMARY:
The goal of this study is to provide an initial pilot test of an Ecological Momentary Intervention (EMI) designed the reduce the distress associated with negative emotion among individuals at risk for suicide that pairs content from a smartphone with a wearable physiological monitor. Participants will be 25 suicidal adult inpatients who will complete three brief therapy sessions with a study therapist and then complete exercises associated with the study for the duration of the inpatient period and for 28 days after they leave the hospital.

DETAILED DESCRIPTION:
The goal of this study is to provide an initial pilot test of an Ecological Momentary Intervention (EMI) designed the reduce the distress associated with negative emotion among individuals at risk for suicide that pairs content from a smartphone with a wearable physiological monitor. Participants will be 25 suicidal adult inpatients who will complete three brief therapy sessions with a study therapist and then complete exercises associated with the study for the duration of the inpatient period and for 28 days after they leave the hospital. During the time they are in the study, participants will be asked to install on their smartphone a mobile application to deliver the therapeutic content and will wear a physiological monitoring device on their wrist (Empatica Embrace) which will monitor objective signals of physiological distress (e.g., skin conductance).

ELIGIBILITY:
Inclusion criteria:

* A recent suicide attempt or serious suicidal ideation (i.e., ideation with at least 70% intent or a suicide plan with access to lethal means),
* The ability to speak and write English fluently, access to an internet-capable smartphone (e.g., an iPhone or Android phone)
* Providing at least one collateral contact in cases where the investigators cannot reach the participant.

Exclusion criteria:

* The presence of any factor that impairs an individual's ability to comprehend and effectively participate in the study including:
* An inability to speak or write English fluently
* The presence of gross cognitive impairment due to florid psychosis, intellectual disability, dementia, or acute intoxication.
* The presence of extremely agitated or violent behavior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in momentary levels of self-reported distress | Through study completion (duration of inpatient stay + 4 weeks post-discharge)
  Assessed via smartphone assessments
Change in momentary levels of physiological distress | Through study completion (duration of inpatient stay + 4 weeks post-discharge)
  Skin conductance (assessed with wearable device)
Change in momentary levels of suicidal thinking | Through study completion (duration of inpatient stay + 4 weeks post-discharge)
  Assessed via smartphone assessments

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kleiman, Principal Investigator — Harvard University
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in accordance with NIH data sharing policies.
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of the completion of the final participant.
Access Criteria: Data will be released to the NIMH's data repository and anyone with access to the repository can access these data.